CLINICAL TRIAL: NCT07246447
Title: Opioid Sparing Anesthesia Using Ketodex Versus Opioid Based Anesthesia in Obese Patients Undergoing Laparoscopic Sleeve Gastrectomy: A Randomized Controlled Trial.
Brief Title: Ketodex Versus Opioid Based Anesthesia in Obese Patients Undergoing Laparoscopic Sleeve Gastrectomy.
Acronym: Ketodex
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mai younes Taha, lecturer of anesthesia , cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ketodex in obesity
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Morbid Obesity
Keywords: ketamine; dexmedatodine; obesity; sleeve gastrectomy
MeSH Terms: conditions — Obesity, Morbid; Obesity | interventions — Ketamine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketodex group (Active Comparator): Group KD: Two syringes containing ketodex-ketamine (1 mg/kg) and dexmedetomidine (1 µg/kg)-each diluted with 0.9% saline and infused over 10 minutes. Maintenance will consist of continuous low-dose infusion of ketamine (0.3 mg/kg/h) and dexmedetomidine (0.5 µg/kg/h) in separate syringes until 15 minutes before the end of surgery.
  Interventions: Drug: ketamine and dexmeditomidine combination
- opioid based group (Active Comparator): Group OP: Two syringes-one containing fentanyl (2 µg/kg) and the other 0.9% saline-infused over 10 minutes. Maintenance will be provided by two continuous saline infusions, prepared to mimic the ketodex infusions, until 15 minutes before the end of surgery.
  Interventions: Drug: Fentanyl (IV)

INTERVENTIONS:
Drug: ketamine and dexmeditomidine combination — Group KD: Two syringes containing ketodex-ketamine (1 mg/kg) and dexmedetomidine (1 µg/kg)-each diluted with 0.9% saline and infused over 10 minutes. Maintenance will consist of continuous low-dose infusion of ketamine (0.3 mg/kg/h) and dexmedetomidine (0.5 µg/kg/h) in separate syringes until 15 minutes before the end of surgery.
  Other Names: ketodex
  Arms: ketodex group
Drug: Fentanyl (IV) — Group OP: Two syringes-one containing fentanyl (2 µg/kg) and the other 0.9% saline-infused over 10 minutes. Maintenance will be provided by two continuous saline infusions, prepared to mimic the ketodex infusions, until 15 minutes before the end of surgery.
  Other Names: opioiod based anesthesia
  Arms: opioid based group

SUMMARY:
comparing Opioid sparing anesthesia using ketodex versus opioid based anesthesia in obese patients undergoing laparoscopic sleeve gastrectomy.

DETAILED DESCRIPTION:
Bariatric surgery has seen a substantial increase, especially among patients with medically complex obesity who struggle to lose weight with traditional approaches . Although advances in anesthetic procedures enhance surgical and clinical outcomes, regular opioid usage in bariatric surgeries might result in adverse effects such as drowsiness, postoperative nausea and vomiting (PONV), respiratory depression, and impaired gastrointestinal motility. These adverse effects increase the risk of postoperative cardiac and respiratory complications .

The key to managing such patients is the utilization of a novel form of anesthesia and analgesia, known as opioid-sparing anesthesia, which has recently been developed to ensure better outcomes . During opioid-sparing anesthesia, the sympathetic nervous system is inhibited by means other than opioid delivery . Such techniques include the use of medications from the alpha-2 agonist group, lidocaine, ketamine, magnesium sulfate, beta-blockers, or gabapentinoids .

Ketamine is an N-methyl-D-aspartate antagonist with analgesic and anti-hyperalgesic properties at low doses . This drug prevents the development of opioid tolerance by minimizing opioid use while reducing postoperative pain, ultimately decreasing opioid-related postoperative morbidity .

Dexmedetomidine, a highly selective α2-adrenoceptor agonist, is used as an adjuvant analgesic in the perioperative period . It improves hemodynamic stability and reduces the stress induced by intubation due to its central sympatholytic action . Furthermore, it decreases the need for opioids and anesthetics, providing additional benefits for obese patients .

By lowering the required dosages, adding a low dose of ketamine to dexmedetomidine is thought to result in less toxicity than using either medication alone . Vishnuraj et al. concluded that the combination of ketamine and dexmedetomidine effectively reduced postoperative opioid consumption; however, their approach involved the use of ketamine as a bolus following induction, in conjunction with a continuous infusion of dexmedetomidine in adults undergoing laparoscopic cholecystectomy .

To the best of our knowledge, the use of both ketamine and dexmedetomidine infusion versus opioid-based anesthesia among patients undergoing bariatric surgery, specifically regarding postoperative pain, has not been previously compared

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years) undergoing Elective Bariatric Surgery .

  * American Society of Anesthesiologists physical status class II or III .
  * body mass index (BMI) > 35 kg/m2 .

Exclusion Criteria:

* • Refusal to participate .

  * Any sensitivity or contraindication to ketamine or dexmedotomidine .
  * Pregnancy or breast feeding .
  * Patients with significant renal impairment .
  * Any patient on regular intake of beta blockers or calcium channel blockers .
  * CNS disorders eg: seizures , raised intra cranial tension .
  * Chronic opioid use.
  * Obese patients with STOP bang score more than 5 .

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Total nalbuphine consumption (mg) during the first 24 hours postoperatively. | during the first 24 hours postoperatively
  Total nalbuphine consumption (mg) during the first 24 hours postoperatively.

SECONDARY OUTCOMES:
Total intraoperative titrated fentanyl dose for each patient. | intraoperative time
Time to extubation, defined as the interval between discontinuation of anesthesia and tracheal extubation | the interval between discontinuation of anesthesia and tracheal extubation
• Time to first postoperative rescue analgesia | during 1st 24 hrs postoperatively.
Postoperative sedation scores. | 1st 24 hours postoperatively
  Sedation assessment: All patients will be monitored postoperatively in the post-anesthesia care unit (PACU) and ward. Sedation will be assessed using the Modified Observer's Assessment of Alertness/Sedation Scale (MOASS) . Scores will be recorded at 0, 10, 30, and 60 minutes from PACU admission.
Postoperative pain scores assessed using the Numerical Rating Scale (NRS). | 1st 24 hours post operatively
  Postoperative pain: Pain will be assessed using the Numerical Rating Scale (NRS, 0 = no pain, 10 = worst pain). Patients will be instructed preoperatively regarding the scale. NRS scores will be recorded at 0, 30, and 60 minutes, and at 2, 6, 12, and 24 hours after surgery.
Postoperative nausea and vomiting (PONV) scores | 1st 24 hours postoperatively
  by using Simplified PONV Impact Scale (SPONVIS) This simplified version, often used for audit and post-discharge review, uses just two main components: Nausea Impact and Vomiting Impact.
  1. Nausea Impact," Based on the patient's assessment of how much the nausea affected their recovery (e.g., ability to eat, walk, or be discharged).","0 to 5 Points (e.g., 0 = No Impact, 5 = Severe Impact/Required hospital stay)"
  2. Vomiting/Retching, Total number of vomiting or retching episodes.,"0 to 5 Points (e.g., 0 = None, 5 = ≥3 episodes)" Total SPONVIS Score Sum of Nausea Impact + Vomiting/Retching Points, Score: 0 to 10 Cut-off for CIPONV Total Score ≥5
Patient satisfaction scores . | during 1st 24 hours postoperatively.
  (0 = not satisfied, 10 = highly satisfied).
Length of hospital stay | 1-2 weeks
  From date of randomization until the date of first documented progression